CLINICAL TRIAL: NCT06050785
Title: Comparison of Infection Rate Between Vancomycin and Gentamycin for Intraoperative Presoaking of Graft in Primary Anterior Cruciate Ligament Reconstruction ( Randomized Controlled Trial )
Brief Title: Infection Rates Between Using of Vancomycin Versus Gentamycin in Primary ACLR
Acronym: ACLR
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Anwer Tawfek, Doctor, Assiut University
Other Study IDs: ACLR
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Vancomycin; Gentamicins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vancomycin group
  Interventions: Drug: Vancomycin
- Gentamycin group
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — ACL graft will be soaked in vancomycin versus gentamycin
  Other Names: Gentamycin

SUMMARY:
The purpose of the study is to compare the efficacy of Vancomycin versus Gentamycin , in reducing infection rates following Anterior Cruciate Ligament Reconstruction .

DETAILED DESCRIPTION:
There has been a marked increase in the number of cases of anterior cruciate ligament reconstruction (ACLR) worldwide. ACLR helps in the restoration of knee instability. But infection following ACLR is a big complication(1) .It may require multiple reoperations in the form of irrigation and debridement, prolonged use of antibiotics, removal of the graft, and sometimes graft revision surgery. It also has increases the risk of early osteoarthritis, and causes graft failure (2,3) .

There are a number of contributing factors that can lead to infection, like the presence of comorbid conditions like diabetes or concomitant open surgical procedures, Use of larger incisions, longer tourniquet time, and use of drain are other contributing factors(4) .Some studies have reported increased chances of infection with hamstring autografts in comparison to patellar tendon autografts and drain application(5,6). The harvested graft is prone to infection from skin flora, and an adequate concentration of antibiotics to inhibit bacterial growth can be achieved with the local application of antibiotics over the graft(7) .The most common pathogen after ACLR is staphylococci, accounting for 90% of cases of septic arthritis (8,9).

Vancomycin is commonly used locally in the surgery in Orthopaedics because of the relative safety for local use in high dosis, and bactericidal action against organisms like Staphylococcus aureus (10) on the other hand there are concerns about its use because of antibiotic resistance, high cost, and graft toxicity(11) . Several studies evaluated the effect of gentamicin solution on ACLR(7). Gentamycin offers an advantage in terms of activity against staphylococci, Gram-negative pathogens, and pseudomonas, along with being cost-effective(7).

The objective of the present study is to compare the infection rate with pre-soaking of harvested grafts in Vancomycin vesus Gentamycin during ACLR.

ELIGIBILITY:
Inclusion Criteria:

* 1) any patient for ACLR

Exclusion Criteria:

* 1) Revision ACL surgery 2) Previous Knee Surgery 3) Associated knee operations other than meniscal surgery (eg.HTO) 4) Open ACL reconstruction 5) Immune suppressed patients (eg. diabetic and patients taking steroids )

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient admitted to Assiut University hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment the infection rates between using the Vancomycin versus Gentamycin | 1-10-2023 to 1-10-2024

SECONDARY OUTCOMES:
Functional outcome and recurrence rate after ACL reconstruction after the use of different antibiotics . Rerupture rate | 1-10-2023 to 1-10-2024

IPD SHARING:
Plan to Share IPD: No